CLINICAL TRIAL: NCT02667184
Title: The Effect of a Low FODMAP Oral Nutrition Supplement On Breath Hydrogen Response In Health Human Subjects
Brief Title: The Effect of a Low FODMAP Oral Nutrition Supplement On Breath Hydrogen Response In Healthy Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1507E75043
Record Dates: First submitted 2016-01-15; First posted 2016-01-28 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low FODMAP Oral Nutrition Supplement 1 (Experimental): Low FODMAP Oral Nutrition Supplement
  Interventions: Dietary Supplement: Low FODMAP Oral Nutrition Supplement
- Low FODMAP Oral Nutrition Supplement 2 (Experimental): Low FODMAP Oral Nutrition Supplement
  Interventions: Dietary Supplement: Low FODMAP Oral Nutrition Supplement
- Low FODMAP Oral Nutrition Supplement 3 (Experimental): Low FODMAP Oral Nutrition Supplement
  Interventions: Dietary Supplement: Low FODMAP Oral Nutrition Supplement
- FOS Supplement (Experimental): Supplement containing fructooligosaccharides
  Interventions: Dietary Supplement: Low FODMAP Oral Nutrition Supplement

INTERVENTIONS:
Dietary Supplement: Low FODMAP Oral Nutrition Supplement

SUMMARY:
The goal of this study is to determine subjective gastrointestinal tolerance response and differences in breath hydrogen response following the consumption of different types of low FODMAP oral nutrition supplements. This randomized, crossover study requires participants to arrive to the lab 12 hours fasted, consume an oral liquid supplement and complete gastrointestinal tolerance questionnaires as well as produce samples for breath hydrogen analysis at various time points over a 4 hour time period.

DETAILED DESCRIPTION:
This randomized, crossover study requires participants to arrive to the lab 12 hours fasted, consume an oral liquid supplement and complete gastrointestinal tolerance questionnaires as well as produce samples for breath hydrogen and methane analysis at various time points over a 4 hour time period. Subjects will also be asked to rate gastrointestinal symptoms via a questionnaire at various time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years with a body mass index between 18-29 kg/m2.
* Demonstrates spoken and written English literacy and able to provide written, informed consent after review of study protocol and procedures.

Exclusion Criteria:

* Use of enemas, proton pump inhibitors, or antibiotics within the past 3 months
* Smoker
* Not a regular breakfast eater
* Self-reported history of a past or current gastrointestinal disease
* High fiber eater (> or = to 3 servings of high fiber foods per day)
* Concurrent or recent (within 30 days) participation in an intervention trial
* Recent weight fluctuations
* Allergies to any of the test products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Breath hydrogen response | baseline
  At baseline, subjects will be asked to exhale a full breath into a sample collection bag. The breath samples will be extracted and measured using the Quintron Breath Track Analyzer. This will be a marker of carbohydrate fermentation in the colon.
Breath hydrogen response | 60 minutes
  At 60 minutes, subjects will be asked to exhale a full breath into a sample collection bag. The breath samples will be extracted and measured using the Quintron Breath Track Analyzer. This will be a marker of carbohydrate fermentation in the colon.
Breath hydrogen response | 120 minutes
  At 120 minutes, subjects will be asked to exhale a full breath into a sample collection bag. The breath samples will be extracted and measured using the Quintron Breath Track Analyzer. This will be a marker of carbohydrate fermentation.
Breath hydrogen response | 240 minutes
  At 240 minutes, subjects will be asked to exhale a full breath into a sample collection bag. The breath samples will be extracted and measured using the Quintron Breath Track Analyzer. This will be a marker of carbohydrate fermentation.

SECONDARY OUTCOMES:
Gastrointestinal tolerance | 48 hours
  Subjects will answer a 7 symptom questionnaire regarding the intensity of gastrointestinal symptoms experienced following consumption of each of the supplements. Questionnaire is adapted from the validated Bovenshen gastrointestinal tolerance questionnaire. Questionnaire is to be completed at baseline, 30 min, 60 min, 90 min, 120 min, 180 min, 12 hours, 24 and 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erickson J, Korczak R, Wang Q, Slavin J. Gastrointestinal tolerance of low FODMAP oral nutrition supplements in healthy human subjects: a randomized controlled trial. Nutr J. 2017 May 25;16(1):35. doi: 10.1186/s12937-017-0256-3. PMID 28545589